CLINICAL TRIAL: NCT07305506
Title: Effects of Post-Match Foam Rolling, Static Stretching, and Passive Rest on Acute Cardiac-Autonomic, Hemodynamic, and Neuromuscular Recovery in National Wrestlers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ali Kamil GÜNGÖR (Other)
Responsible Party: Sponsor-Investigator, Ali Kamil GÜNGÖR, Principal Investigator, Uludag University
Organization: Uludag University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: BUU-WRESTLING-RECOVERY-2025; approval code: 2023-21/18 (Other: Bursa Uludag University Clinical Research Ethics Committee)
Record Dates: First submitted 2025-12-12; First posted 2025-12-26 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Autonomic Function; Hemodynamic Changes; Neuromuscular Adaptations; Exercise and Recovery
Keywords: Wrestling; Recovery; Foam rolling; Static stretching; Passive rest; Heart rate variability; Blood pressure; Anaerobic power; Neuromuscular performance; Countermovement jump; Combat sports; Cardiac autonomic modulation
MeSH Terms: conditions — Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Foam Rolling (Experimental): Participants perform the 9-minute foam rolling recovery protocol immediately after the simulated match.
  Interventions: Procedure: Foam Rolling
- Static Stretching (Experimental): Participants perform the 9-minute static stretching recovery protocol immediately after the simulated match.
  Interventions: Procedure: Static Stretching
- Passive Rest (No Intervention): Participants rest supine for 9 minutes immediately after the simulated match; this serves as a control comparator.

INTERVENTIONS:
Procedure: Foam Rolling — Participants perform a 9-minute foam rolling protocol immediately after the simulated match. Six bilateral muscle groups are targeted: calves, shins, hamstrings, quadriceps, gluteals, and upper back. Each exercise consists of 2 × 30-second rolling per limb, with 30 seconds of rest between exercises and sets. Movements are performed at a metronome-controlled pace (2 seconds up, 2 seconds down). A high-density foam roller (6 × 36 in) is used, and a researcher provides technique supervision throughout.
  Arms: Foam Rolling
Procedure: Static Stretching — Participants perform a 9-minute static stretching routine targeting the same muscle groups as the foam rolling protocol. Each stretch consists of 2 × 30-second holds per limb, with 30 seconds of rest between exercises and sets. Stretches are performed to the point of mild discomfort but without pain. No partner assistance is used, and a researcher supervises to ensure correct technique.
  Arms: Static Stretching

SUMMARY:
This study looks at three common ways athletes recover after a wrestling match: foam rolling, static stretching, and resting. We want to learn which method helps the body recover better in the short time that athletes often have between matches.

Sixteen national-level wrestlers will take part in the study. Each participant will complete all three recovery methods on different days. Before and after each match and recovery session, researchers will measure heart activity, blood pressure, and jump performance. Heart activity is measured through heart rate variability, which shows how well the body's nervous system responds to stress.

The purpose of this study is to find out which recovery method helps the body return to normal faster. The results may help athletes and coaches choose the best recovery strategy during competitions.

DETAILED DESCRIPTION:
This study investigates the acute effects of three practical post-match recovery strategies-foam rolling (FR), static stretching (SS), and passive rest (PR)-on cardiac-autonomic, hemodynamic, and neuromuscular recovery in national-level male wrestlers following a maximal-effort freestyle wrestling match. Wrestling involves high-intensity intermittent actions that substantially elevate cardiovascular and metabolic stress, often requiring athletes to recover rapidly between multiple matches during tournaments. Despite the importance of rapid short-term recovery, limited research has examined accessible, equipment-free recovery methods that can be applied within competition settings.

The study uses a randomized controlled crossover design in which each participant completes all three recovery protocols on separate days. Following a standardized warm-up and a maximal 2×3-min wrestling match, participants perform one of the three 9-min recovery interventions. FR and SS target the same major muscle groups of the lower limbs and upper posterior chain. PR consists of lying supine without movement. Heart rate variability (HRV), blood pressure (BP), and countermovement jump (CMJ) performance are assessed at four time points: pre-match, immediately post-match, immediately post-recovery, and 10 minutes post-recovery.

HRV is recorded using a validated chest-strap heart rate monitor and analyzed with Kubios HRV software to obtain Mean-RR, RMSSD, and SDNN as indicators of cardiac-autonomic modulation. Hemodynamic recovery is evaluated through automated brachial systolic, diastolic, and mean arterial pressure measurements. Neuromuscular recovery is assessed through CMJ height and estimated peak power using an Optojump system and the Sayers equation. All measurements are performed under controlled environmental conditions and standardized protocols.

The study includes national-level freestyle wrestlers with at least five years of competitive experience and no recent injuries or cardiovascular contraindications. A priori power analysis determined that 16 participants provide adequate power (>80%) to detect meaningful differences. All participants complete familiarization before the experimental visits, and all match and recovery protocols follow official wrestling competition procedures.

The primary purpose of this study is to compare whether FR or SS can enhance cardiac-autonomic or hemodynamic recovery relative to PR without compromising neuromuscular performance. Secondary aims include identifying whether either modality facilitates parasympathetic reactivation or BP normalization during the first 10 minutes following completion of the recovery protocol. The findings may inform coaches, sport scientists, and athletes about the practicality and acute effectiveness of common recovery practices used during wrestling tournaments.

ELIGIBILITY:
Inclusion Criteria:

* being freestyle wrestlers,
* holding an active wrestling license for at least 5 years
* possessing at least a C-level National Athlete Certificate (having represented Turkey in at least one international senior wrestling tournament organized by United World Wrestling),
* having trained regularly for the last 12 months,
* having had no injuries in the past 12 months.

Exclusion Criteria:

* having any cardiovascular health issues
* using medications or substances affecting the respiratory or cardiovascular system
* using ergogenic dietary supplements (e.g., creatine, caffeine)
* having a resting systolic blood pressure (SBP) ≥140 mmHg and diastolic blood pressure (DBP) ≥90 mmHg

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2024-02-25 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
RMSSD (root mean square of successive differences) - heart rate variability | Pre-match (baseline), immediately post-match, immediately post-recovery, and 10 minutes post-recovery
  RMSSD will be derived from R-R interval recordings to assess short-term cardiac-parasympathetic modulation and acute autonomic recovery following each post-match recovery intervention.
Mean RR and SDNN - heart rate variability | Pre-match (baseline), immediately post-match, immediately post-recovery, and 10 minutes post-recovery
  Mean RR (average R-R interval) and SDNN (standard deviation of normal R-R intervals) will be calculated from R-R recordings to characterize overall autonomic modulation across time points.

SECONDARY OUTCOMES:
Brachial Blood Pressure (SBP, DBP, MAP) | Pre-match (baseline), immediately post-match, immediately post-recovery, and 10 minutes post-recovery
  Systolic (SBP), diastolic (DBP), and mean arterial pressure (MAP) will be measured using an automated oscillometric device to evaluate hemodynamic recovery after each intervention.
Countermovement Jump (CMJ) height and peak power | Pre-match (baseline), immediately post-match, immediately post-recovery, and 10 minutes post-recovery
  Vertical CMJ height (and derived peak power via Sayers equation) will be measured to assess neuromuscular fatigue and recovery following each post-match recovery method. Two trials performed per time point; best score used.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Kamil Güngör, Phd, Principal Investigator — Uludağ university
Locations (1):
- Bursa Uludağ University, Faculty of Sport Sciences, Bursa, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains sensitive physiological information (e.g., HRV and blood pressure measurements) from a small sample of athletes, which may pose risks to participant privacy even after anonymization. Additionally, institutional policies do not permit external sharing of raw participant-level data. Only aggregated results will be made available upon reasonable request.

REFERENCES:
- [Result] Laborde S, Wanders J, Mosley E, Javelle F. Influence of physical post-exercise recovery techniques on vagally-mediated heart rate variability: A systematic review and meta-analysis. Clin Physiol Funct Imaging. 2024 Jan;44(1):14-35. doi: 10.1111/cpf.12855. Epub 2023 Oct 2. PMID 37754676
- [Result] D'Amico A, Gillis J, McCarthy K, Leftin J, Molloy M, Heim H, Burke C. FOAM ROLLING AND INDICES OF AUTONOMIC RECOVERY FOLLOWING EXERCISE-INDUCED MUSCLE DAMAGE. Int J Sports Phys Ther. 2020 May;15(3):429-440. PMID 32566379
- [Result] Behm DG, Chaouachi A. A review of the acute effects of static and dynamic stretching on performance. Eur J Appl Physiol. 2011 Nov;111(11):2633-51. doi: 10.1007/s00421-011-1879-2. Epub 2011 Mar 4. PMID 21373870
- [Result] Behm DG, Blazevich AJ, Kay AD, McHugh M. Acute effects of muscle stretching on physical performance, range of motion, and injury incidence in healthy active individuals: a systematic review. Appl Physiol Nutr Metab. 2016 Jan;41(1):1-11. doi: 10.1139/apnm-2015-0235. Epub 2015 Dec 8. PMID 26642915
- [Result] Healey KC, Hatfield DL, Blanpied P, Dorfman LR, Riebe D. The effects of myofascial release with foam rolling on performance. J Strength Cond Res. 2014 Jan;28(1):61-8. doi: 10.1519/JSC.0b013e3182956569. PMID 23588488
- [Result] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287
- [Result] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068